CLINICAL TRIAL: NCT06607562
Title: Protective Effect of Probiotics BC99 on Liver Function in Long-Term Alcohol Consumers: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effectiveness and Safety of Probiotics in Protecting Liver Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK2024012
Record Dates: First submitted 2024-09-11; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Experimental): 10B CFU/Sachet/Day BC99 before meals; Storage: Store in cool and dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic group
- Placebo (Placebo Comparator): Maltodextrin one Sachet/Day before meals; Storage: Store in cool and dry place without sun exposure.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Probiotic group — The experimental phase of this study lasted for 56 days, during which we will measure participants' liver function, such as alanine aminotransferase (ALT) at baseline and end.
  Arms: Probiotics group
Dietary Supplement: Placebo group — The experimental phase of this study lasted for 56 days, during which we will measure participants' liver function, such as alanine aminotransferase (ALT) at baseline and end.
  Arms: Placebo

SUMMARY:
To evaluate the effectiveness and safety of using probiotics to protect the liver function of long-term alcohol consumers

ELIGIBILITY:
Inclusion Criteria:

1. A history of long-term heavy alcohol consumption, equivalent to ethanol intake ≥40g/day for over 1 year. The conversion formula is: ethanol (g) = volume of ethanol-containing beverage (mL) × ethanol content (%) × 0.8 (specific gravity of ethanol);
2. Body Mass Index (BMI) between 18kg/m² and 25kg/m²;
3. Voluntarily signed a written informed consent form, agreeing to participate in this study;
4. Agreed to comply with the study protocol and restrictions;
5. Subjects (including male participants) have no plans for conception from 14 days prior to screening until 6 months after the end of the trial and voluntarily agree to use effective contraception.

Exclusion Criteria:

1. Patients with various types of viral hepatitis, autoimmune liver disease, drug-induced liver damage, vascular liver disease, genetic metabolic liver disease, or primary liver cancer;
2. Individuals who have recently consumed substances with similar functions to the tested product, potentially affecting the study results;
3. Patients with severe allergies or immune deficiencies;
4. Pregnant, breastfeeding, or women with plans for pregnancy;
5. Individuals with severe diseases of vital organs such as cardiovascular, pulmonary, hepatic, renal conditions, or those with diabetes, severe thyroid disorders, metabolic diseases, malignant tumors, or severe immune system disorders;
6. Individuals who have used antibiotics within the past two weeks;
7. Participants who did not comply with the required consumption of the tested product or missed follow-ups, making it impossible to evaluate the effectiveness;
8. Other participants deemed unsuitable by the researchers.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
liver function changes | 56 days
  To evaluate its effects on liver function in patients with alcohol-induced liver injury, with a primary focus on alanine aminotransferase (ALT) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wu, Dr., Study Chair — Henan University of Science and Technology
Locations (1):
- Wu Ying, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No